CLINICAL TRIAL: NCT05780138
Title: Implementation of the Parents Taking Action With Caregivers of Young Autistic Children in Paraguay
Brief Title: Implementation of the Parents Taking Action in Paraguay
Acronym: PTA-Paraguay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004046
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Depression; Autism
Keywords: international research; autism; developmental disabilities; caregiver training
MeSH Terms: conditions — Depression; Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Pre-post-test intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will receive 10 remote sessions with the curriculum
  Interventions: Behavioral: Parents Taking Action

INTERVENTIONS:
Behavioral: Parents Taking Action — Educational intervention designed to provide caregivers of children with autism information about autism, and strategies to advocate and support their child's development.

SUMMARY:
The principal aim of this study is to conduct a single group design pilot of a psychoeducational caregiver training (i.e., culturally adapted Parents Taking Action) with a group of family caregivers of young children with autism in Paraguay. The following research questions will be addressed:

Research Question #1: What is the feasibility and acceptability of the intervention? Research Question #2: Do participants improve between pre and post-test on outcome measures? Parents will receive 10 weekly remote sessions on information about autism and strategies to support their child's development. The weekly sessions will be held via telehealth by the researcher and 2 and 2 Paraguayan trained parents of autistic individuals.

DETAILED DESCRIPTION:
The adapted intervention, Parents Taking Action, will consist of 10 weekly online group sessions among family caregivers, the researcher, and 2 Paraguayan trained parents of autistic individuals (Promotoras). The weekly remote sessions will be conducted on a video-chat platform, in Spanish (See Appendix A for curriculum outline).

The promotoras who deliver the sessions will be Paraguayan and will offer the sessions in Spanish. Promotoras will receive 10 hours of training on content and procedures prior to the beginning of the intervention.

Piloting the Intervention The Pilot will consist of a one group pre and post-test design with no control group.

Sample and Recruitment. Twenty family caregivers in Paraguay will be recruited for this pilot study. Primary caregivers are the ones who do most of the care and parenting of the child. Family caregivers will be recruited and will be eligible if (1) they live in Paraguay, (2) are the primary caregivers of a child with autism who is 0-8 years old, and (3) are18 years old or older. All recruitment materials will be in Spanish. Families who express interest in participation will be contacted by a trained research assistant to complete consent forms and to schedule the baseline assessment. After a cohort of 10 to 20 families have been recruited, the pilot intervention will be scheduled.

Data Source/Data Collection. Parents/ family caregivers will complete objective and self-report assessments at baseline and post-intervention follow-up through telephone or videochat interviews with trained students. One interview will be conducted at baseline and one at follow-up to collect the full battery of measures. See Appendix B for a list of the measures. Participants will not receive any compensation to participate in the study. After completing the intervention, family caregivers will be invited to attend an additional individual interview in which we will seek feedback on the social validity of the content and delivery of the intervention. Interviews will be held in Spanish.

Acceptability measures include: (1) Satisfaction with the intervention, which will be evaluated using a survey to be completed by parents/family caregivers after the 10 individual sessions. Satisfaction survey will include questions about accessibility and adequacy of the content; and (2) Optional Social validity interview, which will include questions about the social validity of the goals, the procedures, and the outcomes. Feasibility measures include (1) attendance at individual and family group sessions based on attendance logs; participants who miss sessions will be called to inquire about barriers to attendance; (2) retention at post-intervention; and (3) intervention fidelity checklist. To monitor fidelity, we will utilize self-reported checklists to be completed by the researcher and the promotoras at the end of each session.

Outcome measures:

Family caregivers will complete a total of 4 family caregiver outcome measures. First, Help and support for their child is a 26 item likert-type scale (i.e., not at all/a little/ somewhat/ almost/ completely) which includes questions related to (a) understanding their child's strengths, needs, and abilities, (b) Knowing their rights and advocating for their child, (c) helping their child develop and learn, (d) having support systems, and (e) accessing the community. The second outcome measure is related to family caregivers' depression. This 20-item questionnaire includes questions regarding the family caregiver's feelings during the last week (e.g., happiness, hopefulness, sleep, fearfulness). The third questionnaire is regarding family caregivers' empowerment to use different caregiving strategies with their children. This is an 11-item questionnaire, and family caregivers will mark the degree to which they agree or disagree with the statements. Finally, a 40 item, true or false knowledge questionnaire related to the content presented in the sessions. Additionally, a family caregiver -reported measure will also be included to measure child outcomes. The social communication questionnaire which is a 40-item questionnaire regarding their child's social communication skills and behaviors.

Data Analysis: Descriptive statistics will be used to summarize feasibility and acceptability measures. To generate estimates, we will compute group-specific means and standard deviations for outcome measures. We will use two tailed t-tests to examine differences between baseline and follow-up on outcome measures.

Qualitative data from social validity measures will be video and audio recorded through zoom. A researcher will write a summary of the interview and share it with the participant for member-check. Recordings will be transcribed verbatim in Spanish and translated to English. A bilingual, bicultural member of the research team will review the transcriptions and translations for accuracy. Transcripts will be coded using thematic analysis and deductive coding using the a priori coding scheme that will include (1) social validity of the goals; (2) social validity of the procedures; and (3) social validity of the outcomes. At least two members of the research team will engage in open and deductive coding and will develop a code book, followed by a second round of coding using the codes including in the codebook. At least one of the members of the research team will be bilingual and will refer to the original Spanish transcripts as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Live in Paraguay
2. Be a parent or primary family caregiver
3. Be 18 years old or older
4. Child has a diagnosis of autism
5. Child is between 2 and 8 years old

Exclusion Criteria:

1. Primary Language is not Spanish
2. Does not have access to a device with connection to the internet

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Family Outcome Measure, 24 items, range 0 to 120. Higher better | from baseline to 4 months
  Change from baseline helping and supporting their child at 4 months,
Epidemiological Studies -Depression, 20 items, minimum 0 maximum 60, higher worse. | from baseline to 4 months
  Change from baseline caregivers' depression at 4 months
caregivers' empowerment to use different caregiving strategies, 11 items, 0-44, higher is better | : from baseline to 4 months
  Change from baseline caregivers' depression at 4
Caregiver Knowledge Questionnaire, 40 items, 0-40 higher is better | from baseline to 4 months
  Change from baseline caregivers' knowledge about autism at 4 months.
Social Communication Questionnaire, 40-items, 0-40, higher is worst | from baseline to 4 months
  Change from baseline caregiver -reported social communication questionnaire at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Magana, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Maybe shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after the completion of the study
Access Criteria: Researcher from a recognized institution